CLINICAL TRIAL: NCT03331770
Title: Multicentric Study to Evaluate the Efficacy and Tolerability of an Innovative Formulation of Benzalkonium Chloride-free Latanoprost in Patients With Primary Open-Angle Glaucoma
Brief Title: Efficacy and Tolerability of an Innovative Formulation of BAK-free Latanoprost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Poen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLEMU03
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Primary Open-angle Glaucoma
Keywords: Benzalkonium Chloride; Latanoprost; BAK-free; Glaucoma; Ocular hypertension; conjunctival hyperemia; BUT; OSDI; Schirmer I; Corneal staining; Tear meniscus height
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: A prospective, open-label, single-arm, multicenter, 12-week study
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- BAK-free latanoprost ophthalmic emulsion (Experimental): Patients with primary open-angle glaucoma who were using BAK-containing latanoprost ophthalmic solution for ≥ 6 months (baseline), switched to a new formulation of latanoprost ophthalmic product
  Interventions: Drug: Latanoprost Ophthalmic Product

INTERVENTIONS:
Drug: Latanoprost Ophthalmic Product — Multidose bottle, preserved with potassium sorbate, that can be stored at room temperature up to 30°C during all shelf life, the emulsion does not require shaking before use
  Other Names: Louten® Emulsion

SUMMARY:
This study evaluates the efficacy and tolerability of a new formulation of latanoprost without Benzalkonium Chloride (BAK-free). Patients with open-angle glaucoma who were using BAK-containing latanoprost ophthalmic solution for ≥6 months, switched to BAK-free latanoprost ophthalmic emulsion.

DETAILED DESCRIPTION:
Latanoprost is a prostaglandin F2alfa analogue that increases the uveoscleral outflow of aqueous humor, resulting in a intraocular pressure (IOP) reduction. Benzalkonium chloride (BAK) is usually employed in formulations of prostaglandin analogues due to its dual action of preservative and adjuvant in the formulation. However, this preservative has known toxic effects on the ocular surface, causing ocular dryness and discomfort on long-term use. Benzalkonium Chloride-free (BAK-free)Latanoprost is a new formulation approved for the use in patients with primary open angle glaucoma /ocular hypertension. In this study, patients that were using BAK-containing latanoprost for ≥6 months, switched to a new formulation of BAK-free latanoprost ophthalmic emulsion to evaluate its hypotensive action and quantify the changes in ocular surface parameters.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years
* Diagnosed with primary open-angle glaucoma or pseudoexfoliative glaucoma.
* Receiving containing-BAK latanoprost as monotherapy for at least 6 months
* Pachymetry between 520 and 580 microns
* Informed consent given

Exclusion Criteria:

* History of allergic hypersensitivity or poor tolerance to latanoprost or any components of the formula
* Angle closure glaucoma or secondary glaucoma
* History of recent previous glaucoma surgery or trabeculoplasty (less than 1 year of surgery)
* History of cataract surgery during the last 6 months
* History of uveitis or intraocular inflammation
* Corneal alteration
* Pregnant patients, who wish to conceive or who are in the nursing period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | At the baseline (still on treatment with BAK-containing latanoprost)
  Intraocular pressure (IOP) is the fluid pressure inside the eye. Tonometry is the method eye care professionals use to determine it. IOP is an important aspect in the evaluation of patients at risk from glaucoma. Most tonometers measure pressure in millimeters of mercury (mmHg).
Intraocular pressure | After 4 weeks of treatment with BAK-free latanoprost
  Intraocular pressure (IOP) is the fluid pressure inside the eye. Tonometry is the method eye care professionals use to determine it. IOP is an important aspect in the evaluation of patients at risk from glaucoma. Most tonometers measure pressure in millimeters of mercury (mmHg).
Intraocular pressure | After 8 weeks of treatment with BAK-free latanoprost
  Intraocular pressure (IOP) is the fluid pressure inside the eye. Tonometry is the method eye care professionals use to determine it. IOP is an important aspect in the evaluation of patients at risk from glaucoma. Most tonometers measure pressure in millimeters of mercury (mmHg).
Intraocular pressure | After 12 weeks of treatment with BAK-free latanoprost
  Intraocular pressure (IOP) is the fluid pressure inside the eye. Tonometry is the method eye care professionals use to determine it. IOP is an important aspect in the evaluation of patients at risk from glaucoma. Most tonometers measure pressure in millimeters of mercury (mmHg).

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | At the baseline (still on treatment with BAK-containing latanoprost)
  The OSDI score is a valid and reliable instrument for measuring dry eye disease severity (normal, mild to moderate, and sever) and effect on vision related function. It is determined using OSDI questionnaire (score). The OSDI score is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal patients and patients with dry eye disease.
Ocular Surface Disease Index (OSDI) | After 4 weeks of treatment with BAK-free latanoprost
  The OSDI score is a valid and reliable instrument for measuring dry eye disease severity (normal, mild to moderate, and sever) and effect on vision related function. It is determined using OSDI questionnaire (score). The OSDI score is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal patients and patients with dry eye disease.
Ocular Surface Disease Index (OSDI) | After 8 weeks of treatment with BAK-free latanoprost
  The OSDI score is a valid and reliable instrument for measuring dry eye disease severity (normal, mild to moderate, and sever) and effect on vision related function. It is determined using OSDI questionnaire (score). The OSDI score is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal patients and patients with dry eye disease.
Ocular Surface Disease Index (OSDI) | After 12 weeks of treatment with BAK-free latanoprost
  The OSDI score is a valid and reliable instrument for measuring dry eye disease severity (normal, mild to moderate, and sever) and effect on vision related function. It is determined using OSDI questionnaire (score). The OSDI score is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal patients and patients with dry eye disease.
Conjunctival hyperemia | At the baseline (still on treatment with BAK-containing latanoprost)
  Patients on treatment with prostaglandin analogues preserved with BAK suffer from conjunctival hyperemia. It is the most common side effect that leads to discontinuation or non-compliance. It is determined with the slit lamp. It is classified as patients without hyperemia or with mild, moderate, or severe hyperemia.
Conjunctival hyperemia | After 4 weeks of treatment with BAK-free latanoprost
  Patients on treatment with prostaglandin analogues preserved with BAK suffer from conjunctival hyperemia. It is the most common side effect that leads to discontinuation or non-compliance. It is determined with the slit lamp. It is classified as patients without hyperemia or with mild, moderate, or severe hyperemia.
Conjunctival hyperemia | After 8 weeks of treatment with BAK-free latanoprost
  Patients on treatment with prostaglandin analogues preserved with BAK suffer from conjunctival hyperemia. It is the most common side effect that leads to discontinuation or non-compliance. It is determined with the slit lamp. It is classified as patients without hyperemia or with mild, moderate, or severe hyperemia.
Conjunctival hyperemia | After 12 weeks of treatment with BAK-free latanoprost
  Patients on treatment with prostaglandin analogues preserved with BAK suffer from conjunctival hyperemia. It is the most common side effect that leads to discontinuation or non-compliance. It is determined with the slit lamp. It is classified as patients without hyperemia or with mild, moderate, or severe hyperemia.
Schirmer I test | At the baseline (still on treatment with BAK-containing latanoprost)
  Schirmer test measures the production of tears. This test consists of placing a small strip of filter paper inside the lower eyelid (inferior fornix). The eyes are closed for 5 minutes. The paper is then removed and the amount of moisture is measured (millimeter).
Schirmer I test | After 4 weeks of treatment with BAK-free latanoprost
  Schirmer test measures the production of tears. This test consists of placing a small strip of filter paper inside the lower eyelid (inferior fornix). The eyes are closed for 5 minutes. The paper is then removed and the amount of moisture is measured (millimeter).
Schirmer I test | After 8 weeks of treatment with BAK-free latanoprost
  Schirmer test measures the production of tears. This test consists of placing a small strip of filter paper inside the lower eyelid (inferior fornix). The eyes are closed for 5 minutes. The paper is then removed and the amount of moisture is measured (millimeter).
Schirmer I test | After 12 weeks of treatment with BAK-free latanoprost
  Schirmer test measures the production of tears. This test consists of placing a small strip of filter paper inside the lower eyelid (inferior fornix). The eyes are closed for 5 minutes. The paper is then removed and the amount of moisture is measured (millimeter).
Break up time (BUT) | At the baseline (still on treatment with BAK-containing latanoprost)
  Tear film break-up time (TBUT) is a method for determining the stability of the tear film and checking evaporative dry eye. In testing for TBUT, sodium fluorescein dye is added to the eye and the tear film is observed under the slit lamp while the patient avoids blinking until tiny dry spots develop. The BUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film.
Break up time (BUT) | After 4 weeks of treatment with BAK-free latanoprost
  Tear film break-up time (TBUT) is a method for determining the stability of the tear film and checking evaporative dry eye. In testing for TBUT, sodium fluorescein dye is added to the eye and the tear film is observed under the slit lamp while the patient avoids blinking until tiny dry spots develop. The BUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film.
Break up time (BUT) | After 8 weeks of treatment with BAK-free latanoprost
  Tear film break-up time (TBUT) is a method for determining the stability of the tear film and checking evaporative dry eye. In testing for TBUT, sodium fluorescein dye is added to the eye and the tear film is observed under the slit lamp while the patient avoids blinking until tiny dry spots develop. The BUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film.
Break up time (BUT) | After 12 weeks of treatment with BAK-free latanoprost
  Tear film break-up time (TBUT) is a method for determining the stability of the tear film and checking evaporative dry eye. In testing for TBUT, sodium fluorescein dye is added to the eye and the tear film is observed under the slit lamp while the patient avoids blinking until tiny dry spots develop. The BUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film.
Corneal epithelial fluorescein staining | At the baseline (still on treatment with BAK-containing latanoprost)
  This is a test that uses orange dye (fluorescein) and a blue light to detect damage to the cornea. Fluorescein does not stain intact corneal epithelium but does stain corneal stroma, thus demarcating the area of the epithelial loss. Number of patients with corneal epithelial defects classified as inferior punctata keratitis or central corneal keratitis.
Corneal epithelial fluorescein staining | After 4 weeks of treatment with BAK-free latanoprost
  This is a test that uses orange dye (fluorescein) and a blue light to detect damage to the cornea. Fluorescein does not stain intact corneal epithelium but does stain corneal stroma, thus demarcating the area of the epithelial loss. Number of patients with corneal epithelial defects classified as inferior punctata keratitis or central corneal keratitis.
Corneal epithelial fluorescein staining | After 8 weeks of treatment with BAK-free latanoprost
  This is a test that uses orange dye (fluorescein) and a blue light to detect damage to the cornea. Fluorescein does not stain intact corneal epithelium but does stain corneal stroma, thus demarcating the area of the epithelial loss. Number of patients with corneal epithelial defects classified as inferior punctata keratitis or central corneal keratitis.
Corneal epithelial fluorescein staining | After 12 weeks of treatment with BAK-free latanoprost
  This is a test that uses orange dye (fluorescein) and a blue light to detect damage to the cornea. Fluorescein does not stain intact corneal epithelium but does stain corneal stroma, thus demarcating the area of the epithelial loss. Number of patients with corneal epithelial defects classified as inferior punctata keratitis or central corneal keratitis.
Tear meniscus height | At the baseline (still on treatment with BAK-containing latanoprost)
  The height of the tear meniscus is related to the tear secretion rate and tear stability, and it is a good indicator of the overall tear volume. It is measured with a slit lamp and classified as normal, increased or decreased (millimeter).
Tear meniscus height | After 4 weeks of treatment with BAK-free latanoprost
  The height of the tear meniscus is related to the tear secretion rate and tear stability, and it is a good indicator of the overall tear volume. It is measured with a slit lamp and classified as normal, increased or decreased (millimeter).
Tear meniscus height | After 8 weeks of treatment with BAK-free latanoprost
  The height of the tear meniscus is related to the tear secretion rate and tear stability, and it is a good indicator of the overall tear volume. It is measured with a slit lamp and classified as normal, increased or decreased (millimeter).
Tear meniscus height | After 12 weeks of treatment with BAK-free latanoprost
  The height of the tear meniscus is related to the tear secretion rate and tear stability, and it is a good indicator of the overall tear volume. It is measured with a slit lamp and classified as normal, increased or decreased (millimeter).

CONTACTS AND LOCATIONS:
Overall Officials: Alejo Peyret, PhD, Principal Investigator — Hospital Durand, Argentina; Javier Casiraghi, PhD, Study Chair — Hospital de Clínicas "Jose de San Martin"; Daniel Grigera, PhD, Study Director — Hospital Santa Lucia
Locations (1):
- Laboratoarios Poen, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walimbe T, Chelerkar V, Bhagat P, Joshi A, Raut A. Effect of benzalkonium chloride-free latanoprost ophthalmic solution on ocular surface in patients with glaucoma. Clin Ophthalmol. 2016 May 9;10:821-7. doi: 10.2147/OPTH.S102976. eCollection 2016. PMID 27274186
- [Background] Munoz Negrete FJ, Lemij HG, Erb C. Switching to preservative-free latanoprost: impact on tolerability and patient satisfaction. Clin Ophthalmol. 2017 Mar 21;11:557-566. doi: 10.2147/OPTH.S126042. eCollection 2017. PMID 28356710
- [Background] Cucherat M, Stalmans I, Rouland JF. Relative efficacy and safety of preservative-free latanoprost (T2345) for the treatment of open-angle glaucoma and ocular hypertension: an adjusted Indirect comparison meta-analysis of randomized clinical trials. J Glaucoma. 2014 Jan;23(1):e69-75. doi: 10.1097/IJG.0b013e3182a075e6. PMID 23881267
- [Background] Denis P; Monoprost French Study Group. [Unpreserved latanoprost in the treatment of open-angle glaucoma and ocular hypertension. A multicenter, randomized, controlled study]. J Fr Ophtalmol. 2016 Sep;39(7):622-30. doi: 10.1016/j.jfo.2016.05.006. Epub 2016 Aug 25. French. PMID 27567675
- [Background] Sanford M. Preservative-free latanoprost eye drops in patients with primary open-angle glaucoma/ocular hypertension. Clin Drug Investig. 2014 Jul;34(7):521-8. doi: 10.1007/s40261-014-0203-4. PMID 24895141